CLINICAL TRIAL: NCT01810614
Title: A New Diet for Patients With Autosomal Dominant Polycystic Disease (ADPKD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13493
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD; PKD; Kidney Disease; ADPKD diet
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADPKD Diet (Experimental): All study participants will follow their regular diet for 8 days. After that, they will be asked to follow the ADPKD diet for a total of 4 weeks.
  Interventions: Other: ADPKD Diet

INTERVENTIONS:
Other: ADPKD Diet — Diet specifically designed for people with ADPKD

SUMMARY:
Recent evidence has shown that kidney volume predicts the likelihood of developing renal insufficiency over a finite length of time in ADPKD, suggesting a linkage between the growth of cysts and the harm they do to kidney function. Recent studies indicate that the rate of kidney volume increase is hastened by excess dietary protein, salt, and potential net acid precursors, and slowed by increased water intake sufficient to lower plasma vasopressin levels.

Diets are commonly prescribed to treat ADPKD and other renal patients with disease near the end-stage, but there is currently no specific diet prescription that takes potentially harmful dietary elements into account for ADPKD patients in the earliest stages of the disease. This study will examine a novel diet for ADPKD created by the researcher termed the ADPKD diet.

ELIGIBILITY:
Inclusion Criteria:

* Have not been prescribed dietary restrictions or enhancements
* Blood pressure <135/85 mmHg with or without specific treatment
* Willingness to participate for at least one month
* Diet history consistent with the excretion of >30 mEq NAE / day based on usual dietary intake

Exclusion Criteria:

* Other active diseases requiring pharmacologic agents
* Unstable weight (+/- 2 kg) for 3 months prior to enrollment
* Food allergies
* Pregnancy or lactating
* Confounding medications, i.e. bicarbonate, citrate
* Individuals who do not consume meat for personal, religious, or health reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
ADPKD diet impact on net acid excretion | Change from Baseline to Day 36
  The difference in net acid excretion from a participants regular diet and the ADPKD diet

SECONDARY OUTCOMES:
Acceptance of ADPKD diet | 36 days
  Ease with which diet will be embraced by participants
Kidney injury markers | Change from Baseline to Day 36
  Change in urine markers of renal injury in participants

CONTACTS AND LOCATIONS:
Overall Officials: Debra Sullivan, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Taylor JM, Ptomey L, Hamilton-Reeves JM, Sullivan DK, Creed C, Carlson SE, Wesson DE, Grantham JJ, Gibson CA. Experiences and Perspectives of Polycystic Kidney Disease Patients following a Diet of Reduced Osmoles, Protein, and Acid Precursors Supplemented with Water: A Qualitative Study. PLoS One. 2016 Aug 18;11(8):e0161043. doi: 10.1371/journal.pone.0161043. eCollection 2016. PMID 27537328
- [Derived] Taylor JM, Hamilton-Reeves JM, Sullivan DK, Gibson CA, Creed C, Carlson SE, Wesson DE, Grantham JJ. Diet and polycystic kidney disease: A pilot intervention study. Clin Nutr. 2017 Apr;36(2):458-466. doi: 10.1016/j.clnu.2016.01.003. Epub 2016 Jan 11. PMID 26811129